CLINICAL TRIAL: NCT02127970
Title: A Phase 3b, Double-Blind, Multicenter, Randomized Study to Compare the Efficacy and Safety of Single Dose Dalbavancin to a Two Dose Regimen of Dalbavancin for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Single Dose vs. Two Dose Regimen of Dalbavancin for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUR001-303
Record Dates: First submitted 2014-04-25; First posted 2014-05-01 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Abscess; Wound Infection; Surgical Site Infection; Cellulitis
MeSH Terms: conditions — Abscess; Wound Infection; Surgical Wound Infection; Cellulitis | interventions — dalbavancin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-Dose Dalbavancin (Experimental): Single-dose of dalbavancin 1500 mg intravenous (IV) infusion over 30 minutes on Day 1 followed by dalbavancin-matching placebo IV infusion over 30 minutes on Day 8 for participants with creatinine clearance (CrCl) ≥30 mL/min or with CrCl <30 mL/min who were receiving regular hemodialysis or peritoneal dialysis. For participants with CrCl <30 mL/min who were not receiving regular hemodialysis or peritoneal dialysis, the dalbavancin dose was 1000 mg.
  Interventions: Drug: Dalbavancin; Drug: Dalbavancin-matching Placebo
- Two-Dose Dalbavancin (Experimental): Two-dose regimen of dalbavancin 1000 mg IV infusion over 30 minutes on Day 1 followed by 500 mg IV infusion over 30 minutes on Day 8 for participants with CrCl ≥30 mL/min or with CrCl <30 mL/min who were receiving regular hemodialysis or peritoneal dialysis. For participants with CrCl <30 mL/min who were not receiving regular hemodialysis or peritoneal dialysis, the dalbavancin doses were 750 mg on Day 1 and 375 mg on Day 8.
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin IV infusion over 30 minutes.
  Other Names: DALVANCE®
Drug: Dalbavancin-matching Placebo — Dalbavancin-matching placebo IV infusion over 30 minutes.
  Arms: Single-Dose Dalbavancin

SUMMARY:
To compare the efficacy of treatment with a single dose of dalbavancin 1500 mg to treatment with a two dose regimen of dalbavancin (1000 mg on Day 1 followed by 500 mg on Day 8) in participants with known or suspected Gram-positive acute bacterial skin and skin structure infections (ABSSSI) at 48 -72 hours after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 - 85 years of age.
* Signed and dated informed consent document.
* Major abscess, surgical site infection, traumatic wound infection or cellulitis suspected or confirmed to be caused by Gram-positive bacteria.
* At least two (2) local signs and symptoms of acute bacterial skin and skin structure infection (ABSSSI and at least one systemic sign of infection.
* Participant willing and able to comply with study procedures.

Exclusion Criteria:

* A contra-indication to dalbavancin.
* Pregnant or nursing females.
* Sustained shock.
* Participation in another study of an investigational drug or device within 30 days.
* Receipt of a systemically or topically administered antibiotic with a Gram-positive spectrum that achieves therapeutic concentrations in the serum or at the site of the ABSSSI within 14 days prior to randomization. An exception is allowed for participants receiving a single dose of a short-acting (half-life ≤ 12 hours) antibacterial drug prior to randomization; up to 25% of participants may have received such therapy.
* Infection due to an organism known prior to study entry to be resistant to dalbavancin or vancomycin (vancomycin MIC (minimum inhibitory concentration) >8 μg/mL).
* Evidence of meningitis, necrotizing fasciitis, gas gangrene, gangrene, septic arthritis, osteomyelitis; endovascular infection, such as clinical and/or echocardiographic evidence of endocarditis or septic thrombophlebitis.
* Infections caused exclusively by Gram-negative bacteria (without Gram-positive bacteria present) and infections caused by fungi, whether alone or in combination with a bacterial pathogen.
* Venous catheter entry site infection.
* Infections involving a diabetic foot ulceration, perirectal abscess or a decubitus ulcer.
* Participant with an infected device, even if the device is removed. Examples include infection of: prosthetic cardiac valve, vascular graft, a pacemaker battery pack, joint prosthesis, hemodialysis catheter, implantable pacemaker or defibrillator, intra-aortic balloon pump, left ventricular assist device, a peritoneal dialysis catheter, or a neurosurgical device such as a ventricular peritoneal shunt, intra-cranial pressure monitor, or epidural catheter.
* Gram-negative bacteremia, even in the presence of Gram-positive infection or Gram-positive bacteremia. Note: If a Gram-negative bacteremia develops during the study, or is subsequently found to have been present at Baseline, the participant should be removed from study treatment and receive appropriate antibiotic(s) to treat the Gram-negative bacteremia. Such participants must have an end of treatment (EOT) visit performed within 3 calendar days after discontinuing study medication but are required to have AEs (adverse events) reported through the Final Visit.
* Participants whose ABSSSI is the result of having sustained full or partial thickness burns.
* Participants with an infection involving a limb with evidence of critical ischemia of an affected limb defined as any of the following criteria: absent or abnormal Doppler wave forms, toe blood pressure of <45 mm Hg, ankle brachial index <0.5, and/ or critical ischemia as assessed by a vascular surgeon.
* Participants with ABSSSI such as superficial/simple cellulitis/erysipelas, impetiginous lesion, furuncle, or simple abscess that only requires surgical drainage for cure.
* Concomitant condition requiring any antibiotic therapy that would interfere with the assessment of study drug for the condition under study.
* Anticipated need of antibiotic therapy for longer than 14 days.
* Participants who are placed in a hyperbaric chamber as adjunctive therapy for the ABSSSI.
* More than 2 surgical interventions (defined as procedures conducted under sterile technique and typically unable to be performed at the bedside) for the ABSSSI, or participants who are expected to require more than 2 such interventions.
* Medical conditions in which chronic inflammation may preclude assessment of clinical response to therapy even after successful treatment (e.g., chronic stasis dermatitis of the lower extremity).
* Absolute neutrophil count <500 cells/mm^3.
* Known or suspected human immunodeficiency virus (HIV) infected participants with a CD4 (cluster of differentiation 4) cell count <200 cells/mm3 or with a past or current acquired immunodeficiency syndrome (AIDS)-defining condition and unknown CD4 count.
* Participants with a recent bone marrow transplant (in post-transplant hospital stay).
* Participants receiving oral steroids >20 mg prednisolone per day (or equivalent) or receiving immunosuppressant drugs after organ transplantation.
* Participants with a rapidly fatal illness, who are not expected to survive for 3 months.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participants inappropriate for entry into this study.
* Prior participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2014-04-18 (Actual); Primary Completion 2015-03-11 (Actual); Study Completion 2015-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — Allergan
Locations (78):
- United States (25):
  - 110, Montgomery, Alabama
  - 103, Anaheim, California
  - 117, Long Beach, California
  - 106, Long Beach, California
  - 118, Modesto, California
  - 104, San Diego, California
  - 113, San Diego, California
  - 115, San Diego, California
  - 116, San Diego, California
  - 108, Stockton, California
  - 105, Sylmar, California
  - 112, Washington D.C., District of Columbia
  - 107, Orlando, Florida
  - 120, Saint Cloud, Florida
  - 114, Augusta, Georgia
  - 122, Columbus, Georgia
  - 125, Savannah, Georgia
  - 119, Eunice, Louisiana
  - 101, Springfield, Massachusetts
  - 109, Detroit, Michigan
  - 121, Butte, Montana
  - 123, Omaha, Nebraska
  - 111, Toledo, Ohio
  - 126, Franklin, Tennessee
  - 127, Smyrna, Tennessee
- Bulgaria (3):
  - 802, Sofia
  - 800, Sofia
  - 801, Sofia
- Croatia (2):
  - 200, Zagreb
  - 201, Zagreb
- Estonia (3):
  - 253, Tallinn
  - 252, Tallinn
  - 251, Tartu
- Georgia (4):
  - 302, Kutaisi
  - 303, Tbilisi
  - 300, Tbilisi
  - 301, Tbilisi
- Hungary (4):
  - 352, Debrecen
  - 353, Kaposvár
  - 354, Pécs
  - 351, Szeged
- Latvia (5):
  - 402, Daugavpils
  - 401, Liepāja
  - 403, Rēzekne
  - 400, Riga
  - 404, Riga
- Romania (4):
  - 501, Cluj-Napoca, Cluj
  - 502, Bucharest
  - 500, Bucharest
  - 503, Bucharest
- Russia (7):
  - 555, Vsevolozhsk, Leningradskaya Oblast'
  - 557, Irkutsk
  - 552, Moscow
  - 554, Moscow
  - 553, Novosibirsk
  - 551, Saint Petersburg
  - 556, Tomsk
- Serbia (4):
  - 600, Belgrade
  - 601, Belgrade
  - 603, Niš
  - 602, Novi Sad
- South Africa (10):
  - 756, Breyten
  - 760, Cape Town
  - 752, Dundee
  - 755, Johannesburg
  - 751, Middleburg
  - 758, Port Elizabeth
  - 757, Pretoria
  - 753, Pretoria
  - 759, Pretoria
  - 754, Worcester
- Ukraine (7):
  - 700, Cherkasy
  - 704, Dnipropetrovsk
  - 706, Ivano-Frankivsk
  - 701, Ivano-Frankivsk
  - 705, Kharkiv
  - 703, Lviv
  - 702, Zaporizhzhya

REFERENCES:
- [Derived] Gonzalez PL, Rappo U, Akinapelli K, McGregor JS, Puttagunta S, Dunne MW. Outcomes in Patients with Staphylococcus aureus Bacteremia Treated with Dalbavancin in Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):423-434. doi: 10.1007/s40121-021-00568-7. Epub 2021 Dec 14. PMID 34905144
- [Derived] Rappo U, Gonzalez PL, Puttagunta S, Akinapelli K, Keyloun K, Gillard P, Liu Y, Dunne MW. Single-dose dalbavancin and patient satisfaction in an outpatient setting in the treatment of acute bacterial skin and skin structure infections. J Glob Antimicrob Resist. 2019 Jun;17:60-65. doi: 10.1016/j.jgar.2019.02.007. Epub 2019 Feb 20. PMID 30797084
- [Derived] Dunne MW, Puttagunta S, Giordano P, Krievins D, Zelasky M, Baldassarre J. A Randomized Clinical Trial of Single-Dose Versus Weekly Dalbavancin for Treatment of Acute Bacterial Skin and Skin Structure Infection. Clin Infect Dis. 2016 Mar 1;62(5):545-51. doi: 10.1093/cid/civ982. Epub 2015 Nov 26. PMID 26611777

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 698 participants were randomly assigned in a 1:1 ratio to the following treatment groups: Single-dose dalbavancin group, received a single dose of dalbavancin intravenous (IV) on Day 1, and a matching placebo IV on Day 8; Two-dose dalbavancin group, received dalbavancin IV on Day 1 and Day 8.
Period: Overall Study
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Started | 349 | 349
Completed | 323 | 322
Not Completed | 26 | 27
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 14 | 14
Not completed — Reason not Specified | 4 | 7
Not completed — Pregnancy | 0 | 1
Not completed — Subject Withdrew Consent | 5 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin | Total
Number analyzed (Participants) | 349 | 349 | 698
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (14.83) | 48.3 (14.74) | 48.2 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 146 | 291
  Male | 204 | 203 | 407

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Clinical Responders 48-72 Hours After the Initiation of Study Drug
Description: Clinical responder was defined as a participant who was alive and had received no rescue therapy for acute bacterial skin and skin structure infection (ABSSSI) prior to the 48-72 hour infection site assessment (if an antibiotic has been given for another reason, the participant will not be considered a non-responder for this reason); and examination of the participant's ABSSSI lesion demonstrates a decrease of ≥ 20% in lesion area (calculated as the longest length multiplied by the longest perpendicular width) relative to the baseline measurement.
Time Frame: Up to 48-72 hours after the initiation of study drug
Population: ITT Population included all randomized participants regardless of whether or not they received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 349 | 349
percentage of participants | 81.4 | 84.2
Statistical Analysis 1: Comparison: Single-Dose Dalbavancin vs Two-Dose Dalbavancin; Test type: Non-Inferiority — The non-inferiority hypothesis test was to be a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the 95% CI for the difference in responder rates is greater than -10%, then the single-dose dalbavancin regimen was to be declared non-inferior to the two dose dalbavancin regimen; Difference = -2.9, 95% CI 2-sided [-8.5 to 2.8] — For the difference in clinical responder rates (single-dose group minus two dose group), the 95% CI was calculated using the Miettinen and Nurminen method without adjustment

2. Secondary Outcome: Percentage of Participants by Clinical Status at End of Treatment (EOT) and Final Visit (FV)
Description: Clinical Success is defined as follows: For evaluation at EOT visit, lesion area must be decreased by ≥80% from baseline and at FV lesion area must be decreased by ≥90% from baseline; Temperature is ≤37.6°C; Local signs of tenderness to palpation and swelling/induration are no worse than mild; For evaluation at EOT visit, local signs of fluctuance and localized heat/warmth must be improved from baseline and no worse than mild, and at FV local signs of fluctuance and localized heat/warmth must be absent; for participants with a wound infection the severity of purulent drainage is improved and no worse than mild relative to baseline. Clinical Failure is defined as the opposite to success or if the participant died during the study period up to visit or received study therapy for ABSSSI beyond the protocol treatment period. Clinical status is Indeterminate if any of the data needed to determine clinical success or clinical failure were missing.
Time Frame: End of Treatment (Day 14-15 after the initiation of study drug) and Final Visit (28 ±2 days after the initiation of study drug)
Population: ITT Population included all randomized participants regardless of whether or not they received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 349 | 349
percentage of participants
  EOT; Clinical Success | 84.0 | 84.8
  EOT; Clinical Failure | 12.0 | 10.3
  EOT; Indeterminate | 4.0 | 4.9
  FV; Clinical Success | 84.5 | 85.1
  FV; Clinical Failure | 8.0 | 7.2
  FV; Indeterminate | 7.4 | 7.3

3. Other Pre Specified Outcome: Percentage of Participants by Clinical Status Based on Localized Fluctuance and Heat/Warmth at End of Treatment (EOT)
Description: Clinical Success was defined as localized fluctuance and heat/warmth that if present at Baseline must be improved and no worse than mild. Clinical Failure was defined as the opposite to success. Clinical status was Indeterminate if any of the data needed to determine clinical success or clinical failure were missing.
Time Frame: EOT (Day 14-15)
Population: ITT Population included all randomized participants regardless of whether or not they received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 349 | 349
percentage of participants
  Clinical Success | 84.8 | 85.4
  Clinical Failure | 7.7 | 6.9
  Indeterminate | 7.4 | 7.7

4. Other Pre Specified Outcome: Percentage of Participants by Investigator Assessment of Clinical Outcome
Description: A successful outcome was based on resolution or improvement of all signs and symptoms of the infection to such an extent that no further antibacterial treatment was given. An unsuccessful outcome was the opposite of successful. An Indeterminate outcome was defined as any of the data needed to determine a successful or unsuccessful outcome were missing.
Time Frame: Day 3-4, Day 8, EOT (Day 14-15) and Final Visit (Day 28 +/- 2 days)
Population: ITT Population included all randomized participants regardless of whether or not they received study drug. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 347 | 344
percentage of participants
  Successful Outcome (Day 3-4) | 93.4 | 93.0
  Unsuccessful Outcome (Day 3-4) | 0.3 | 0.9
  Indeterminate (Day 3-4) | 6.3 | 6.1
  Successful Outcome (Day 8) | 92.2 | 93.3
  Unsuccessful Outcome (Day 8) | 0.6 | 0.3
  Indeterminate (Day 8) | 7.2 | 6.4
  Successful Outcome (EOT) | 92.5 | 92.7
  Unsuccessful Outcome (EOT) | 2.9 | 1.5
  Indeterminate (EOT) | 4.6 | 5.8
  Successful Outcome (Final Visit) | 90.2 | 91.0
  Unsuccessful Outcome (Final Visit) | 2.6 | 1.7
  Indeterminate (Final Visit) | 7.2 | 7.3

5. Other Pre Specified Outcome: Percentage of Participants Achieving Clinical Outcome of Success Based on Key Target Pathogen at Baseline
Description: A successful outcome was based on resolution or improvement of all signs and symptoms of the infection to such an extent that no further antibacterial treatment was given.
Time Frame: Day 3-4 and EOT (Day 14-15)
Population: Microbiological Intent-to-treat (MicroITT) Population included all ITT participants who had at least 1 Gram-positive bacterial pathogen isolated at Baseline. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 210 | 220
percentage of participants
  Staphylococcus aureus (Day 3-4): number analyzed (Participants) | 139 | 156
  Staphylococcus aureus (Day 3-4) | 88.5 | 85.3
  Streptococcus agalactiae (Day 3-4): number analyzed (Participants) | 6 | 6
  Streptococcus agalactiae (Day 3-4) | 100.0 | 66.7
  Streptococcus anginosus group (Day 3-4): number analyzed (Participants) | 33 | 19
  Streptococcus anginosus group (Day 3-4) | 93.9 | 100.0
  Streptococcus dysgalactiae (Day 3-4): number analyzed (Participants) | 4 | 3
  Streptococcus dysgalactiae (Day 3-4) | 100.0 | 100.0
  Streptococcus pyogenes (Day 3-4): number analyzed (Participants) | 14 | 22
  Streptococcus pyogenes (Day 3-4) | 100.0 | 81.8
  Enterococcus faecalis (Day 3-4): number analyzed (Participants) | 4 | 10
  Enterococcus faecalis (Day 3-4) | 100.0 | 80.0
  Staphylococcus aureus (EOT): number analyzed (Participants) | 139 | 156
  Staphylococcus aureus (EOT) | 87.8 | 91.7
  Streptococcus agalactiae (EOT): number analyzed (Participants) | 6 | 6
  Streptococcus agalactiae (EOT) | 83.3 | 83.3
  Streptococcus anginosus group (EOT): number analyzed (Participants) | 33 | 19
  Streptococcus anginosus group (EOT) | 81.8 | 89.5
  Streptococcus dysgalactiae (EOT): number analyzed (Participants) | 4 | 3
  Streptococcus dysgalactiae (EOT) | 100.0 | 100.0
  Streptococcus pyogenes (EOT): number analyzed (Participants) | 14 | 22
  Streptococcus pyogenes (EOT) | 92.9 | 81.8
  Enterococcus faecalis (EOT): number analyzed (Participants) | 4 | 10
  Enterococcus faecalis (EOT) | 100.0 | 100.0

6. Other Pre Specified Outcome: Percentage of Participants With Complete Resolution of Local Signs of Infection
Description: Resolution of Local Signs of Infection that include absence of purulence/drainage, erythema, heat/localized warmth, pain/tenderness to palpation, fluctuance, and swelling/induration.
Time Frame: Day 3-4, Day 8, EOT (Day 14-15) and Final Visit (Day 28 +/- 2 days)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 349 | 349
percentage of participants
  Day 3-4: number analyzed (Participants) | 321 | 324
  Day 3-4 | 1.9 | 1.5
  Day 8: number analyzed (Participants) | 328 | 329
  Day 8 | 22.3 | 21.1
  EOT Visit: number analyzed (Participants) | 334 | 338
  EOT Visit | 56.3 | 56.2
  Final Visit: number analyzed (Participants) | 295 | 295
  Final Visit | 85.8 | 89.8

7. Other Pre Specified Outcome: Change From Baseline in Participant's Assessment of Pain
Description: Using the Brief Pain Inventory Scale, participants rated their pain "right now" on a scale where: 0=no pain to 10=pain as bad as you can imagine. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) to Day 3-4, Day 8, EOT (Day 14-15) and Final Visit (Day 28 + /- 2 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 349 | 349
Scores on a scale
  Baseline | 7.7 (2.09) | 7.8 (2.12)
  Change from Baseline to Day 3-4 | -3.9 (2.46) | -3.8 (2.43)
  Change from Baseline to Day 8 | -5.9 (2.53) | -5.8 (2.68)
  Change from Baseline to EOT Visit | -6.9 (2.37) | -6.9 (2.53)
  Change from Baseline to Final Visit | -7.5 (2.19) | -7.4 (2.40)

8. Other Pre Specified Outcome: Percentage of Participants by Resource Utilization Categories
Description: Resource Utilization Categories included: Any additional visits (including urgent care), Any additional procedures, Any additional tests, Any home visits or nursing care and Any ER Visits. The percentage of participants in each category is reported.
Time Frame: Final Visit (Day 28 +/- 2 days)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 323 | 322
percentage of participants
  Any Additional Visits (including Urgent Care) | 1.2 | 0.6
  Any Additional Procedures | 1.5 | 1.6
  Any Additional Tests | 1.9 | 2.8
  Any Home Visits or Home Nursing Care | 1.5 | 1.2
  Any ER Visits | 0.3 | 0.9

9. Other Pre Specified Outcome: Percentage of Participants by Skin and Soft Tissue Infection-Convenience (SSTI-C) Questionnaire: Overall Satisfaction Response
Description: The SSTI-C Questionnaire is an 11-item self-reported questionnaire that measures subjective experiences of the participant. One of the items assessed was overall satisfaction with treatment. Participants answered the question: "Overall, how satisfied were you with your antibiotic treatment?" using one of the following responses: Extremely satisfied, Moderately satisfied, Not at all satisfied, Slightly satisfied and Very satisfied. The percentage of participants in each category is reported.
Time Frame: EOT (Day 14-15)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
Number analyzed (Participants) | 338 | 332
percentage of participants
  Extremely Satisfied | 53.6 | 56.9
  Moderately Satisfied | 9.5 | 7.2
  Not at all Satisfied | 0.9 | 0.9
  Slightly Satisfied | 0.3 | 0.9
  Very Satisfied | 35.8 | 33.7

ADVERSE EVENTS:
Time Frame: Up to 28 Days
Description: The number of participants at risk for Serious Adverse Events and Adverse Events was based on the Safety Population that included all participants who received at least 1 dose of study treatment.
Arm/Group | Single-Dose Dalbavancin | Two-Dose Dalbavancin
All-Cause Mortality (participants affected / at risk) | 1/349 | 1/346
Serious Adverse Events (participants affected / at risk) | 7/349 | 5/346
Other Adverse Events (participants affected / at risk) | 0/349 | 0/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Dose Dalbavancin (N=349) | Two-Dose Dalbavancin (N=346)
Vitreous haemorrhage (Eye disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that the first results publication shall be made in conjunction with a joint multi-center publication. If the multi-center publication is not submitted within 18 months after conclusion of the study at all sites, or if the sponsor confirms not to publish the results, the PI may publish the results from the institution subject to terms of the clinical trial agreement. The publication must be sent to Sponsor at least 60 days before the intended submission date for reference and comment.